CLINICAL TRIAL: NCT00503581
Title: A Randomized Phase II Evaluation of Continuous Progestin Therapy vs. Sequential Progestin Therapy in the Treatment of Endometrial Intraepithelial Neoplasia (EIN) From a Referred Cohort of Atypical Endometrial Hyperplasia (AEH) or EIN Patients That Desire Uterine Preservation
Brief Title: Megestrol in Treating Patients With Endometrial Neoplasia or Endometrial Hyperplasia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0224; NCI-2009-00594 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0224; CDR0000555427; GOG-0224 (Other: Gynecologic Oncology Group); GOG-0224 (Other: DCP); GOG-0224 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: High Grade Squamous Intraepithelial Neoplasia; Stage 0 Uterine Corpus Cancer
MeSH Terms: conditions — Squamous Intraepithelial Lesions | interventions — Biopsy; Megestrol Acetate

ARMS (3):
- Regimen 1 (megestrol acetate, surgery) (Experimental): Patients receive oral megestrol twice daily every day for 24 weeks. Approximately twelve weeks after treatment starts, clinical blood tests are obtained and research serum and plasma collected. Twenty-four weeks constitutes one course of treatment and a pill count is performed during the 12-week f/u visit and at the completion of the treatment course to determine compliance. After progestin therapy the patient has an induced-withdrawal bleed. Patients in this arm undergo a re-evaluation biopsy and hysterectomy a minimum of two weeks and a maximum of eight weeks after completing the megestrol treatment.
  Interventions: Procedure: Biopsy; Other: Laboratory Biomarker Analysis; Drug: Megestrol Acetate; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery
- Regimen 2 (megestrol acetate, surgery) (Experimental): Patients receive oral megestrol twice daily for two weeks continuously followed by no treatment for two weeks. This course is repeated for a total of 24 weeks. Approximately twelve weeks after treatment starts, clinical blood tests are obtained and research serum and plasma collected. Twenty-four weeks constitutes one course of treatment and a pill count is performed during the 12-week f/u visit and at the completion of the treatment course to determine compliance. After progestin therapy the patient has an induced-withdrawal bleed. Patients in this arm undergo a re-evaluation biopsy and hysterectomy a minimum of two weeks and a maximum of eight weeks after the megestrol treatment.
  Interventions: Procedure: Biopsy; Other: Laboratory Biomarker Analysis; Drug: Megestrol Acetate; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery
- Regimen 3 (surgery/biopsy) (Active Comparator): (Closed as of 6/3/2010) Patients do not receive megestrol. At the discretion of the managing physician, patients undergo the re-evaluation biopsy and hysterectomy anytime between 2-20 weeks after enrollment and randomization.
  Interventions: Procedure: Biopsy; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: Bx
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Megestrol Acetate — given orally
  Other Names: 17-Hydroxy-6-methylpregna-4,6-diene-3,20-dione acetate; 17.alpha.-Acetoxy-6-methylpregna-4,6-diene-3,20-dione; 6-Dehydro-6-methyl-17.alpha.-acetoxyprogesterone; 6-Methyl-6-dehydro-17.alpha.-acetoxyprogesterone; BDH 1298; BDH-1298; Maygace; Megace; Megestat; Megestil; Niagestin; Ovaban; Pallace; SC-10363
  Arms: Regimen 1 (megestrol acetate, surgery); Regimen 2 (megestrol acetate, surgery)
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Therapeutic Conventional Surgery — undergo hysterectomy

SUMMARY:
This randomized phase II trial is studying how well megestrol works in treating patients with endometrial neoplasia or endometrial hyperplasia. Estrogen can cause the growth of endometrial cancer cells. Hormone therapy using megestrol may fight endometrial cancer by blocking the use of estrogen by the abnormal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the frequency of complete remission by a central pathology review panel in diagnosed endometrial intraepithelial neoplasia (EIN) patients treated for 24 weeks with oral continuous versus interrupted progestin therapy.

SECONDARY OBJECTIVES:

I. To evaluate whether quality of life is superior in patients who take continuous megestrol versus sequential megestrol by evaluating mood, concerns about weight changes and bleeding.

TERTIARY:

I. To assess the expression levels of PTEN using immunohistochemistry and to explore the association of PTEN expression levels with patient response to treatment.

II. To assess the expression levels of the hormone receptors ER and PR using immunohistochemistry and to explore the association of ER/PR expression levels with patient response to treatment.

III. To assess histomorphometry and karyometry characteristics of the pre-treatment biopsy in this patient population.

IV. To identify patterns of protein and glycoprotein expression associated with invasive cancer in serum specimens obtained from patients with a diagnosis of atypical endometrial hyperplasia (AEH) or EIN.

V. To assess differences in plasma concentrations of megestrol acetate HPLC in this patient population.

VI. To assess patient compliance to their treatment regimen using HPLC.

OUTLINE: Patients are stratified according to the collection method of the initial/intake biopsy (dilatation and curettage vs all other methods). Patients are randomized to 1 of the following treatment regimens:

REGIMEN 1: Patients receive oral megestrol twice daily every day for 24 weeks. Approximately twelve weeks after treatment starts, clinical blood tests are obtained and research serum and plasma collected. Twenty-four weeks constitutes one course of treatment and a pill count is performed during the 12-week f/u visit and at the completion of the treatment course to determine compliance. After progestin therapy the patient has an induced-withdrawal bleed. Patients in this arm undergo a re-evaluation biopsy and hysterectomy a minimum of two weeks and a maximum of eight weeks after completing the megestrol treatment.

REGIMEN 2: Patients receive oral megestrol twice daily for two weeks continuously followed by no treatment for two weeks. This course is repeated for a total of 24 weeks. Approximately twelve weeks after treatment starts, clinical blood tests are obtained and research serum and plasma collected. Twenty-four weeks constitutes one course of treatment and a pill count is performed during the 12-week f/u visit and at the completion of the treatment course to determine compliance. After progestin therapy the patient has an induced-withdrawal bleed. Patients in this arm undergo a re-evaluation biopsy and hysterectomy a minimum of two weeks and a maximum of eight weeks after the megestrol treatment.

REGIMEN 3: (Closed as of 6/3/2010) Patients do not receive megestrol. At the discretion of the managing physician, patients undergo the re-evaluation biopsy and hysterectomy anytime between 2-20 weeks after enrollment and randomization. Patients undergo biopsy and blood sample collection periodically for immunological and pharmacodynamic studies. Samples are analyzed for presence or absence of myoinvasion or deep myoinvasion in hysterectomy specimens, hormone receptivity status, and to compare PTEN status against treatment via karyometry or morphometry, expression of VEGF and tenascin-C (TN-C) via ELISA, presence of TN-C fragmentation via western immunoblots, additional biomarkers via proteomic analysis, protein and glycoprotein expression patterns via electrophoresis and image analysis, and plasma megestrol concentrations via high-performance liquid chromatography (HPLC). Patients complete the Hospital Anxiety and Depression Scale (HADS) and two items on bleeding and weight gain at baseline and periodically during study. A Treatment Decision Assessment is completed at baseline, and for patients withdrawing from the study, a Study Withdraw Assessment is also completed. There will be no additional follow-up on this study after the patient's hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of atypical endometrial hyperplasia (AEH) or endometrial intraepithelial neoplasia (EIN) diagnosed by dilatation and curettage (D&C), Novak curettage, Vabra aspirate, or Pipelle endometrial biopsy at the enrolling institution within 12 weeks of enrollment
* Patients must desire uterine retention for duration of study (18 months or after 3rd biopsy) if they remain EIN negative (-); patients are allowed to attempt pregnancy after their initial post-treatment biopsy without it being a major protocol violation
* Patients must have a GOG performance status of 0, 1, or 2
* White blood cell (WBC) >= 3000
* Platelets >= 100,000
* Granulocytes >= 1,500
* Creatinine =< 2
* Bilirubin =< 1.5 x institutional upper limit normal
* Serum glutamic oxaloacetic transaminase (SGOT) =< 3 x institutional upper limit normal
* Alkaline phosphatase =< 3 x institutional upper limit normal
* Patients of child-bearing potential must have a negative serum pregnancy test prior to starting study drug and prior to each biopsy if capable of becoming pregnant (and at the discretion of the referring physician)
* Patients of childbearing potential must use appropriate non-hormonal contraception while on study medication
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients with a GOG performance status of 3 or 4
* Patients with recognized endometrial carcinoma
* Patients with current or prior history of breast cancer
* Patients with invasive malignancies, with the exception of nonmelanoma skin cancer who had (or have) any evidence of the other cancer present within the past 5 years or whose previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor are excluded
* Patients who are pregnant or lactating
* Patients with a history of thrombophlebitis, thromboembolic phenomena, or cerebrovascular disorders within the past 5 years
* Patients under 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-07; Primary Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Method, Principal Investigator — Gynecologic Oncology Group
Locations (50):
- United States (50):
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Hartford Hospital, Hartford, Connecticut
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Memorial University Medical Center, Savannah, Georgia
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium CCOP, South Bend, Indiana
  - Michiana Hematology Oncology-PC Westville, Westville, Indiana
  - Gynecologic Oncology of West Michigan PLLC, Grand Rapids, Michigan
  - Michiana Hematology Oncology PC-Niles, Niles, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Ozark Health Ventures LLC-Cancer Research for The Ozarks Springfield, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Mount Carmel Health Center West, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates-Midtown, Tulsa, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regimen 1 (Megestrol Acetate, Surgery) | Regimen 2 (Megestrol Acetate, Surgery) | Regimen 3 (Surgery/Biopsy)
Started | 3 | 4 | 2
Completed | 0 | 0 | 0
Not Completed | 3 | 4 | 2
Not completed — Study closed | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Population: Participants enrolled in study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen 1 (Megestrol Acetate, Surgery) | Regimen 2 (Megestrol Acetate, Surgery) | Regimen 3 (Surgery/Biopsy) | Total
Number analyzed (Participants) | 3 | 4 | 2 | 9
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 1 | 2 | 0 | 3
  40-49 years | 0 | 0 | 1 | 1
  50-59 years | 2 | 1 | 0 | 3
  60-69 years | 0 | 1 | 0 | 1
  70-79 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 9
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experience a Response as Determined by a Central Blinded Review of the Three Post Treatment Endometrial
Description: Treated and eligible participants. This study had 0 participants that completed treatment, therefore no analysis was done. Study closed prior to completion. Central blinded review was not performed for any participants in the study.
Time Frame: Up to 12 months after completion of treatment
Population: Treated and eligible participants. There were none.
Arm/Group | Regimen 1 (Megestrol Acetate, Surgery) | Regimen 2 (Megestrol Acetate, Surgery) | Regimen 3 (Surgery/Biopsy)
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change in Quality of Life (QOL) Evaluated Using the Hospital Anxiety and Depression Scale (HADS) and the Two Items on Bleeding and Weight Gain
Description: Eligible and Treated patients. This study had 0 participants that completed study.
Time Frame: Baseline to up to 12 months
Population: Eligible and treated patients. This study was closed before subjects could complete evaluation.
Arm/Group | Regimen 1 (Megestrol Acetate, Surgery) | Regimen 2 (Megestrol Acetate, Surgery) | Regimen 3 (Surgery/Biopsy)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months
Description: All Enrolled subjects.
Arm/Group | Regimen 1 (Megestrol Acetate, Surgery) | Regimen 2 (Megestrol Acetate, Surgery) | Regimen 3 (Surgery/Biopsy)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 2/4 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 (Megestrol Acetate, Surgery) (N=3) | Regimen 2 (Megestrol Acetate, Surgery) (N=4) | Regimen 3 (Surgery/Biopsy) (N=2)
Weight Gain (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 0
Hemorrhage, Gu - Vagina (Vascular disorders) | 0 | 1 | 0
Hemorrhage, Gu - Uterus (Vascular disorders) | 0 | 1 | 0
Edema: Limb (Blood and lymphatic system disorders) | 1 | 0 | 0
Mood Alteration - Anxiety (Nervous system disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less